CLINICAL TRIAL: NCT03469739
Title: Types of Intimate Partner Violence and Women's Health: Findings From the WHO Multi-country Study on Women's Health and Intimate Partner Violence
Brief Title: Types of Intimate Partner Violence and Women's Health
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: UoB2646
Record Dates: First submitted 2016-06-10; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-01

CONDITIONS: Domestic Violence
Keywords: Intimate Partner Violence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study uses data from 29,990 women from 12 different countries collected by the WHO multi-country study on women's health and domestic violence to capture the effect of different types, frequency and timing of IPV on self-reported health, symptoms and suicidal behaviours.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) has detrimental effects on physical and mental health, risks to children and is associated with wider societal and healthcare costs. Previous analysis of the WHO multi-country study on women's health and domestic violence found significant associations between physical and sexual IPV and self-reported ill-health, symptomatology and suicidal behaviours.

Real experience of IPV can comprise different combinations of emotional, physical and sexual abuse, and different timings and frequencies of these. A more nuanced testing of exposure to these different combinations of IPV and associations with health is needed.

This study uses data from 29,990 women from 12 different countries collected by the WHO multi-country study on women's health and domestic violence to capture the effect of different combination types, frequency and timing of IPV on self-reported health, symptoms and suicidal behaviours.

ELIGIBILITY:
Inclusion Criteria:

* The WHO report that in most sites, a representative sample of women was obtained using a two-stage cluster sampling scheme to select households and then only one woman per household was randomly selected per household for interview.

Exclusion Criteria:

-

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study consists of further analysis of 29,990 interviews conducted with women in 12 different countries coordinated by the World Health Organisation. They report in most sites around 1500 women between 15 and 49 years old were interviewed. Countries included were Bangladesh, Brazil, Cambodia, Ethiopia, Japan, Maldives, Namibia, Peru, Samoa, Serbia and Montenegro, Thailand and the United Republic of Tanzania.
Sampling Method: Non-Probability Sample
Enrollment: 29990 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Participant description of their current overall state of health | Preceding 4 weeks
  Participant description of their current overall state of health- a choice of options- excellent, good, fair, poor or very poor.

SECONDARY OUTCOMES:
Participant reported health in the last 4 weeks- problems walking around, doing usual activities, pain or discomfort, problems with memory or concentration, dizziness or vaginal discharge. Measured by questionnaire. | Preceding 4 weeks
  Participant rating of various health aspects in last 4 weeks
Emotional distress. Measured by questionnaire of 20 different symptoms of emotional distress. SRQ-20 (score of 20 different symptoms of emotional distress with yes/no answers) | Preceding 4 weeks
  Self Reporting Questionnaire-20 (SRQ-20)- aggregate score of 20 different symptoms of emotional distress with yes/no answers
Participant reported ever suicidal thoughts or attempts; measured by questionnaire. | Up to 49 years
  Participants reporting ever having suicidal thoughts or ever attempting suicide
Participant reported medication used for sleep/ pain; measured by questionnaire. | Preceding 4 weeks
  Participants reporting medication use

CONTACTS AND LOCATIONS:
Overall Officials: Gene Feder, MD FRCGP, Study Director — University of Bristol; Lucy C Potter, MB ChB, Principal Investigator — University of Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellsberg M, Jansen HA, Heise L, Watts CH, Garcia-Moreno C; WHO Multi-country Study on Women's Health and Domestic Violence against Women Study Team. Intimate partner violence and women's physical and mental health in the WHO multi-country study on women's health and domestic violence: an observational study. Lancet. 2008 Apr 5;371(9619):1165-72. doi: 10.1016/S0140-6736(08)60522-X. PMID 18395577
- [Background] Garcia-Moreno C, Jansen HA, Ellsberg M, Heise L, Watts CH; WHO Multi-country Study on Women's Health and Domestic Violence against Women Study Team. Prevalence of intimate partner violence: findings from the WHO multi-country study on women's health and domestic violence. Lancet. 2006 Oct 7;368(9543):1260-9. doi: 10.1016/S0140-6736(06)69523-8. PMID 17027732